CLINICAL TRIAL: NCT00416286
Title: Phase 1: To Evaluate the Antibacterial Efficacy of Sustained Release Cetylpyridinium Chloride Varnish in Orthodontic Patients
Brief Title: Effect of Sustained-Release Cetylpyridinium Chloride Varnish on Streptococcus Mutans and Lactobacillus in Orthodontic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: 26-23.12.05-HMO-CTIL; 26-23.12.05; code: 1371
Record Dates: First submitted 2006-12-25; First posted 2006-12-27 (Estimated); Last update posted 2006-12-27 (Estimated); Status verified 2006-12

CONDITIONS: Healthy
Keywords: Cetylpyridinium chlorid; Sustained release; orthodontic patients; streptococcus mutans; Lactobacillus; Rate of bacterial load in saliva of orthodontic patients

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of the study is to was to evaluate the anti bacterial efficacy of sustain-release Cetylpyridinium chloride varnish on orthodontic patients.

ELIGIBILITY:
Exclusion Criteria:

* Children under 12y old

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Doron Harari, DMD, Principal Investigator — Orthodontic department, Dental school Hadassah Ein Kerem